CLINICAL TRIAL: NCT02632539
Title: Air-impingement Manipulation to Clear Subglottic Secretion to Prevent Ventilator Associated Pneumonia in Prolonged Intubated Patients：a Randomized Controlled Trial
Brief Title: Air-impingement Manipulation to Clear Subglottic Secretion to Prevent VAP in Prolonged Intubated Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Jiwei LI, RRT-NPS, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJCYH-RCCM-01
Record Dates: First submitted 2015-08-14; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: ventilator associated pneumonia; Subglottic Secretion Drainage; manual air-impingement operation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- subglottic secretion drainage (Active Comparator): The conventional method which we use subglottic secretion drainage to clear subglottic secretion
  Interventions: Procedure: subglottic secretion drainage
- Manual air-impingement operation (Experimental): A method which we invented to clear subglottic secretion
  Interventions: Procedure: Manual air-impingement operation

INTERVENTIONS:
Procedure: Manual air-impingement operation — A method which we invented to clear subglottic secretion
  Arms: Manual air-impingement operation
Procedure: subglottic secretion drainage — The conventional method which we use subglottic secretion drainage to clear subglottic secretion
  Arms: subglottic secretion drainage

SUMMARY:
Ventilator-associated pneumonia (VAP) is the most frequent infection occurring in patients who are admitted to the ICU. The accumulation of respiratory secretions in the subglottic space is a well-proven cause of VAP. Investigators invented a manual method with high-flow air produced by resuscitator to impinge secretion from the subglottic space to oral cavity. Investigators want to compare it with conventional method which uses a special intubation tube with an independent dorsal lumen to suction subglottic secretion.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is the most frequent infection occurring in patients who are admitted to the ICU. The accumulation of respiratory secretions in the subglottic space is a well-proven cause of VAP. Therefore, prevention should include the aspiration of secretions from the subglottic space. Investigators invented a manual method with high-flow air produced by resuscitator to impinge secretion from the subglottic space to oral cavity. This method has been granted as a patent by Chinese national intellectual property patent office, it has been used in investigators' daily work for more than 10 years and more than 20 Chinese ICUs have used it everyday. Investigators want to compare it with conventional method which uses a special intubation tube with an independent dorsal lumen to suction subglottic secretion.

ELIGIBILITY:
Inclusion Criteria:Should meet all the criteria:

* Intubation less than 24 hours before admitting respiratory intensive care unit;
* Anticipated intubation for more than 72 hours;
* Anticipated survival time is more than 2 weeks

Exclusion Criteria:Meet any of these criteria:

* PEEP≥10cmH2O or FiO2≥0.8;
* unstable hemodynamics;
* severe bulla and pneumothorax;
* enrolled in other study;
* cuff leak test is positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with ventilator-associated pneumonia | Up to 28 days

SECONDARY OUTCOMES:
Percentage of participants with ventilator-associated event | Up to 28 days
ICU mortality | Participants will be followed for the duration of ICU stay, an expected average of 4 weeks

OTHER OUTCOMES:
Invasive ventilation duration | Participants will be followed for the duration of invasive ventilation, an expected average of 7-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jiwei Li, Principal Investigator — Beijing Chao Yang Hospital

REFERENCES:
- [Result] Grossman RF, Fein A. Evidence-based assessment of diagnostic tests for ventilator-associated pneumonia. Executive summary. Chest. 2000 Apr;117(4 Suppl 2):177S-181S. doi: 10.1378/chest.117.4_suppl_2.177s. No abstract available. PMID 10816031
- [Result] Damas P, Frippiat F, Ancion A, Canivet JL, Lambermont B, Layios N, Massion P, Morimont P, Nys M, Piret S, Lancellotti P, Wiesen P, D'orio V, Samalea N, Ledoux D. Prevention of ventilator-associated pneumonia and ventilator-associated conditions: a randomized controlled trial with subglottic secretion suctioning. Crit Care Med. 2015 Jan;43(1):22-30. doi: 10.1097/CCM.0000000000000674. PMID 25343570
- [Result] Klompas M. Ventilator-associated pneumonia: is zero possible? Clin Infect Dis. 2010 Nov 15;51(10):1123-6. doi: 10.1086/656738. Epub 2010 Oct 11. No abstract available. PMID 20936977
- [Result] Frost SA, Azeem A, Alexandrou E, Tam V, Murphy JK, Hunt L, O'Regan W, Hillman KM. Subglottic secretion drainage for preventing ventilator associated pneumonia: a meta-analysis. Aust Crit Care. 2013 Nov;26(4):180-8. doi: 10.1016/j.aucc.2013.03.003. Epub 2013 Apr 11. PMID 23583261
- [Result] Ramirez P, Bassi GL, Torres A. Measures to prevent nosocomial infections during mechanical ventilation. Curr Opin Crit Care. 2012 Feb;18(1):86-92. doi: 10.1097/MCC.0b013e32834ef3ff. PMID 22186217
- [Result] Suys E, Nieboer K, Stiers W, De Regt J, Huyghens L, Spapen H. Intermittent subglottic secretion drainage may cause tracheal damage in patients with few oropharyngeal secretions. Intensive Crit Care Nurs. 2013 Dec;29(6):317-20. doi: 10.1016/j.iccn.2013.02.007. Epub 2013 May 31. PMID 23727136
- [Result] Lorente L, Lecuona M, Jimenez A, Mora ML, Sierra A. Influence of an endotracheal tube with polyurethane cuff and subglottic secretion drainage on pneumonia. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1079-83. doi: 10.1164/rccm.200705-761OC. Epub 2007 Sep 13. PMID 17872488
- [Result] Tao Z, Zhao S, Yang G, Wang L, Zhu S. [Effect of two methods of subglottic secretion drainage on the incidence of ventilator-associated pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2014 Apr;37(4):283-6. Chinese. PMID 24969718
- [Result] Bouza E, Perez MJ, Munoz P, Rincon C, Barrio JM, Hortal J. Continuous aspiration of subglottic secretions in the prevention of ventilator-associated pneumonia in the postoperative period of major heart surgery. Chest. 2008 Nov;134(5):938-946. doi: 10.1378/chest.08-0103. Epub 2008 Jul 18. PMID 18641114
- See also: Evidence-based assessment of diagnostic tests for ventilator-associated pneumonia.Executive summary — http://journal.publications.chestnet.org.proxy1.lib.uwo.ca/data/Journals/CHEST/21944/177S.pdf
- See also: Prevention of ventilator-associated pneumonia and ventilator-associated conditions: a randomized controlled trial with subglottic secretion suctioning. — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/25343570
- See also: Ventilator-associated pneumonia: is zero possible? — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/20936977
- See also: Subglottic secretion drainage for preventing ventilator associated pneumonia: a meta-analysis. — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/23583261
- See also: Measures to prevent nosocomial infections during mechanical ventilation. — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/22186217
- See also: Intermittent subglottic secretion drainage may cause tracheal damage in patients with few oropharyngeal secretions. — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/?term=Intermittent+subglottic+secretion+drainage+may+cause+tracheal+damage+in+patients+with+few+oropharyngeal+secretions
- See also: Influence of an endotracheal tube with polyurethane cuff and subglottic secretion drainage on pneumonia. — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/?term=Influence+of+an+endotracheal+tube+with+polyurethane+cuff+and+subglottic+secretion+drainage+on+pneumonia.
- See also: Effect of two methods of subglottic secretion drainage on the incidence of ventilator-associated pneumonia — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/?term=Effect+of+tow+methods+of+subglottic+secretion+drainage+on+the+incidence+of+ventilator-associated+pneumonia.
- See also: Continuous aspiration of subglottic secretions in the prevention of ventilator-associated pneumonia in the postoperative period of major heart surgery. — http://www-ncbi-nlm-nih-gov.proxy1.lib.uwo.ca/pubmed/?term=Continuous+aspiration+of+subglottic+secretions+in+the+prevention+of+ventilator-associated+pneumonia+in+the+postoperative+period+of+major+heart+surgery.